CLINICAL TRIAL: NCT04242290
Title: Is it Possible to Distinguish Cervicogenic Headache From Neck Pain With Cervicospinal Posture?: A Single-blind, Prospective Cross-sectional Trial
Brief Title: Cervicospinal Posture and Pain in Cervicogenic Headache
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Yeliz Bahar Ozdemir, Medical Doctor, Hitit University
Other Study IDs: 19-KAEK-064
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cervicogenic Headache; Neck Pain
Keywords: Cervicogenic headache; Disability; Pain
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervicogenic headache: The group with cervicogenic headaches
  Interventions: Diagnostic Test: Lateral radiography
- Neck pain: The group with isolated neck pain
  Interventions: Diagnostic Test: Lateral radiography

INTERVENTIONS:
Diagnostic Test: Lateral radiography — The lordosis angles were measured on the lateral cervical graphs of all patients.

SUMMARY:
Cervicogenic headache (CEH) is a type of symptomatic headache that is characterized by chronic unilateral headache secondary to cervical spine dysfunction. Generally, it gets worse by neck movements, continuous placement of the head in an awkward position and exposure to external pressure on the upper cervical or occipital region.

The pain was demonstrated to originate from lower cervical disc prolapse and spinal nerve roots in some studies, while it is suggested in some others to occur due to the upper cervical region as well. Although disturbed cervical alignment has been determined in tension headache and migraine, there are few studies with controversial results in the literature investigating the effects of the change in cervical lordosis on CEH. These contradictory results strongly influence the decision of whether exercise should be added to the treatment protocol in CEH and also the creation of an appropriate treatment program by the clinicians. In light of this background, the aim of this study was to compare the cervical radiographs of patients with CEH and patients with neck pain without a headache.

DETAILED DESCRIPTION:
The general demographics, pain status and cervical radiological evaluations of the patients was performed in this prospective, cross-sectional, single-blind study evaluating two different disease groups compatible in age and gender and the two groups were compared.

For inclusion in the Cervicogenic Headache group, inclusion criteria determined by the Cervicogenic Headache International Study Group (CHISG) were used.

Symptoms of all patients were questioned in detail and physical examinations were performed. After obtaining demographic information such as age, height and weight, severity and duration of pain were asked to the patients and Neck Disability Index (NDI) and Visual Analogue Scale (VAS) were used for pain assessment Cervical radiographic analysis was evaluated measuring general cervical lordosis and upper cervical lordosis on lateral standing X-rays using Surgimap®. General cervical lordosis and Upper cervical lordosis measurements were performed on the lateral cervical graph.

ELIGIBILITY:
Inclusion Criteria:

For Cervicogenic headache group

* Unilateral headache, starting from the upper neck/occipital region and spreading to the oculofrontotemporal area on the symptomatic side
* Pain triggered by neck movements and/or continuous awkward positions
* Decreased joint range of motion in the cervical vertebra

Exclusion Criteria:

For Cervicogenic headache group

* Previously diagnosed to have any other syndromes of headache (Migraine, Tension headache, etc.)
* Presence of bilateral headache; For the neck pain group,
* Presence of 2 or more neurological symptoms (decreased upper extremity muscle strength, decreased reflexes and hypoesthesia compatible with the dermatome regions)
* Suggesting nerve root compression (radiculopathy, plexopathy); for both groups,
* Presence of any signs suspicious of central nervous system involvement (hyperreflexia, nystagmus, decreased vision, etc)
* Reluctance to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: It was included 45 women with cervicogenic headaches with an age of 18-50 years and 45 women with only neck pain in the same ages who presented to the Neurosurgery outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
General cervical lordosis | 3 months
  General cervical lordosis is basically measured by the "Cobb" method. In the lateral graph, the angle between the two lines drawn perpendicular to the lines passing on the inferior end plate of the C2 and C7 vertebrae is considered as the "General cervical lordosis angle".

SECONDARY OUTCOMES:
Upper cervical lordosis | 3 months
  For the measurement of upper cervical lordosis, a line is drawn from the uppermost posterior point of the odontoid process to the lowermost posterior point of C2. The second line is drawn to pass between the lowermost-posterior portions of the C3 and C4 cervical vertebrae. The angle between these two lines is considered the "upper cervical lordosis angle"

OTHER OUTCOMES:
Neck disability index | 3 months
  The NDI is the most widely used questionnaire to investigate the disability associated with neck pain.
Visual analog scale | 3 months
  The VAS pain scale is used to measure and monitor pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Bahar Ozdemir, Principal Investigator — Hitit University Erol Olcok Training and Research Hospital
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Farmer PK, Snodgrass SJ, Buxton AJ, Rivett DA. An investigation of cervical spinal posture in cervicogenic headache. Phys Ther. 2015 Feb;95(2):212-22. doi: 10.2522/ptj.20140073. Epub 2014 Oct 9. PMID 25301967
- [Result] Knackstedt H, Krakenes J, Bansevicius D, Russell MB. Magnetic resonance imaging of craniovertebral structures: clinical significance in cervicogenic headaches. J Headache Pain. 2012 Jan;13(1):39-44. doi: 10.1007/s10194-011-0387-4. Epub 2011 Sep 27. PMID 21947945